CLINICAL TRIAL: NCT07256561
Title: Antimicrobial and Anti-inflammatory Effects of Simvastatin as an Intracanal Medication in Endodontically Retreated Teeth With Periapical Radiolucency, Randomized Controlled Clinical Trial
Brief Title: Antimicrobial and Anti-inflammatory Effects of Simvastatin as an Intracanal Medication
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hadeer Maher Mostafa Mohamed (Other Government)
Responsible Party: Sponsor-Investigator, Hadeer Maher Mostafa Mohamed, Assistant Lecturer of Endodontics at Suez University, Faculty of Dental Medicine for Girls
Organization: Faculty of Dental Medicine for Girls (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Effects of Simvastatin
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-08

CONDITIONS: Endodontically Retard Teeth; Periapical Radiolucency
MeSH Terms: interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simvastatin Group (Active Comparator): About 27 Patients will take Simvastatin 10mg tablets which will be crushed into fine particles and dissolved to prepare an intracanal medication with specific concentration according to the antimicrobial sensitivity study.
  Interventions: Procedure: Simvastatin as an intracanal medication
- Calcium hydroxide (Active Comparator): About 27 Patients will be injected by Calcium hydroxide intracanal medication in endodontic retreatment of single rooted teeth with periapical radiolucency.
  Interventions: Procedure: Simvastatin as an intracanal medication

INTERVENTIONS:
Procedure: Simvastatin as an intracanal medication — to evaluate the antimicrobial and anti-inflammatory effects of Simvastatin as an intracanal medication in endodontic retreatment of single rooted teeth with periapical radiolucency.
  Other Names: calcium hydroxide intracanal medication

SUMMARY:
Successful endodontic treatment and a predictable outcome can only be achieved by effective root canal debridement, irrigation, and elimination of microorganisms .

The outcome of endodontic treatment performed in controlled clinical environment has demonstrated success rate around 90%.

In certain cases, endodontic treatment may fail, one of the most common reasons is inability to eliminate microorganisms from the root canal. When non-surgical root canal therapy fails, the treatment options include orthograde re-treatment, periradicular surgery, or extraction.

Simvastatin (SIM) is a drug used primarily to treat hyperlipidemia and protect against cardiovascular diseases. It has been shown to possess pleiotropic effects such as antimicrobial, anti-inflammatory, immunomodulatory, antioxidant, and bone-forming properties .

The side chain of this material has a single methyl group. It inhibits hydroxymethyl glutarylcoenzyme reductase that prevents endogenous cholesterol synthesis

DETAILED DESCRIPTION:
It has been reported that the inflamed/infected periodontal/endodontic content influence cytokines release . These inflammatory mediators, such as interleukin (IL)-1β, tumor necrosis factor α (TNF-α), and prostaglandin E2 (PGE2), have been detected in periapical tissues and root canal exudates .

Proinflammatory cytokines are able to stimulate, either directly or indirectly, the release of matrix metalloproteinases (MMPs) in the periapical/periodontal region, maintaining a persistent inflammatory process. MMPs are deeply involved in the pathogenesis of pulp, periodontal, and periapical tissue destruction.

As a Gram-positive, facultative anaerobe, Enterococcus Faecalis (E. Faecalis) can survive root canal treatment . It can form biofilms and survive prolonged periods of nutritional deprivation. It can also resist acidic and basic conditions and is hard to eradicate .

E. Faecalis is responsible for 20-70% of endodontic failures and secondary endodontic infections . Due to biofilm development and the organism's physicochemical characteristics, which enable it to alter the prevailing environmental and nutritional conditions, it can even thrive in constrained environments .

Accumulated evidence indicates that the tissue destruction in endodontic and periodontal infections is due to host-derived cytokines induced by lipopolysaccharides (LPS/endotoxins), acting as the major components of the outer leaflet of the outer membrane of gram-negative bacteria.

Calcium hydroxide (Ca (OH)2) has been widely used as an intracanal medicament for retreatment of such failed cases, due to its high pH, its ability to stimulate mineralization, its antibacterial properties, and its tissue-dissolving capability .

Hydroxyl ions create free radicals that destroy components of bacterial cell membranes. These free radicals react with bacterial DNA inhibiting DNA replication and cell activity, and cause mutations. Also, the alkaline pH of calcium hydroxide alters enzyme activity, disrupting cellular metabolism and structural proteins .

Simvastatin enhances alkaline phosphatase activity and mineralization and increases the expression of bone sialoprotein, osteocalcin, and type I collagen, and it is shown to have an anti-inflammatory effect by decreasing the production of interleukin-6 and interleukin-8. SIM is reported to stimulate vascular endothelial growth factor (VEGF) release in a dose dependent manner, and the authors of a previous study suggested that statins may promote osteoblast differentiation and bone nodule formation by stimulating VEGF expression in bone tissue.

Simvastatin is also a renowned safe and affordable medication. It is a novel medicinal substance that is still undergoing dental research . Various animal and clinical studies showed that SIM assists in bone regeneration as well as the anti-inflammatory effect when delivered or applied locally.

Periapical radiography is an essential resource in endodontic diagnosis because it offers important evidence on the progression, regression, and persistence of apical periodontitis (AP) . It is known that periapical radiolucency might not be visible radiographically, although they exist clinically. Conventional radiographs used for the management of endodontic problems yield limited information because of the two-dimensional (2D) nature of the images produced, geometric distortion and anatomical noise.

ELIGIBILITY:
Inclusion Criteria:

* Patients had anon contributory medical history.
* Patients of age categories between 20 to 40 years old, with no physical disability or psychological problems.
* Single rooted teeth with type I root canal anatomy.
* Symptomatic cases of failed endodontic treatment with radiographic evidence of periapical bone loss, and the lesion size ranging from 2mm up to 8mm.

Exclusion Criteria:

* Patients with known sensitivity to the pharmaceutical used in this trial
* Patients with former endodontic mishaps (as ledges, transportations, perforations or separated instruments)
* Non restorable teeth
* Presence of an associated sinus tract.
* Advanced periodontal involvement
* Teeth representing root fracture.
* Pregnant women

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-08-10 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-10 (Estimated)

PRIMARY OUTCOMES:
Simvastatin antimicrobial effect | 6 Months
  Following the treatment, patients will be asked to evaluate The antimicrobial effect of Simvastatin intracanal medication

SECONDARY OUTCOMES:
Simvastatin anti-inflammatory effect | 6 Months
  Following the treatment, patients will be asked to evaluate The anti-inflammatory effect of Simvastatin intracanal medication and periapical radiolucency healing.

CONTACTS AND LOCATIONS:
Overall Officials: Mervat Ibrahim Fawzy, Professor, Study Chair — Faculty of Dental Medicine for Girls Al Azhar University
Locations (1):
- Faculty of Dental Medicine for Girls, Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided